CLINICAL TRIAL: NCT00001740
Title: Evaluation of Left Ventricular Volumes by Real-Time 3-Dimensional Echocardiography
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980016; 98-H-0016
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Heart Diseases
Keywords: Cardiac; Function; MRI; Reconstruction; Ultrasound; Heart Disease (Cardiovascular Disease)
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases

SUMMARY:
Quantitative measurements of left ventricular volume and ejection fraction are useful in the management of patients with heart disease. Several imaging methods exist, but are limited by cost, invasiveness, or exposure to radio-isotopes. Conventional echocardiography is a noninvasive method that allows estimation of left ventricular size and function; however, quantitative measurements of volume are not widely used due to lack of reproducibility and inaccurate measurements. Real-time three-dimensional echocardiography is a new technique that can be used to derive volume measurements from a single image acquisition. We hypothesize that real-time three-dimensional echocardiography is an accurate method for making left ventricular volume measurements. We therefore propose to measure left ventricular volumes using real-time three-dimensional echocardiography in human subjects and correlate these measurements with magnetic resonance imaging, a more accurate noninvasive method for obtaining these measurements.

DETAILED DESCRIPTION:
Quantitative measurements of left ventricular volume and ejection fraction are useful in the management of patients with heart disease. Several imaging methods exist, but are limited by cost, invasiveness, or exposure to radio-isotopes. Conventional echocardiography is a noninvasive method that allows estimation of left ventricular size and function; however, quantitative measurements of volume are not widely used due to lack of reproducibility and inaccurate measurements. Real-time three-dimensional echocardiography is a new technique that can be used to derive volume measurements from a single image acquisition. We hypothesize that real-time three-dimensional echocardiography is an accurate method for making left ventricular volume measurements. We therefore propose to measure left ventricular volumes using real-time three-dimensional echocardiography in human subjects and correlate these measurements with magnetic resonance imaging, a more accurate noninvasive method for obtaining these measurements.

ELIGIBILITY:
Normal volunteers and patients with any form of heart disease who agree to undergo MRI and echocardiographic examination studies.

Adults older than the age of 18 years.

No pregnancy, atrial fibrillation, unstable angina, recent myocardial infarction (less than 5 days), or other acute medical illness.

No pacemaker, aneurysm clip, neural stimulator, ear implant, and metallic foreign body such as shrapnel or bullets.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 1997-10; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Siu SC, Levine RA, Rivera JM, Xie SW, Lethor JP, Handschumacher MD, Weyman AE, Picard MH. Three-dimensional echocardiography improves noninvasive assessment of left ventricular volume and performance. Am Heart J. 1995 Oct;130(4):812-22. doi: 10.1016/0002-8703(95)90082-9. PMID 7572591
- [Background] Schroder KM, Sapin PM, King DL, Smith MD, DeMaria AN. Three-dimensional echocardiographic volume computation: in vitro comparison to standard two-dimensional echocardiography. J Am Soc Echocardiogr. 1993 Sep-Oct;6(5):467-75. doi: 10.1016/s0894-7317(14)80465-3. PMID 8260164